CLINICAL TRIAL: NCT00518284
Title: A Phase II Trial of ABI-007 (Paclitaxel Albumin-bound Particles) for the Prevention of Restenosis Following Revascularization of the Superficial Femoral Artery (SFA)
Brief Title: Prevention of Restenosis Following Revascularization
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to changing sponsor priorities, and was not based on safety or outcomes data.
Sponsor: Celgene Corporation (Industry)
Responsible Party: Sponsor
Organization: Celgene (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CVR002
Record Dates: First submitted 2007-08-16; First posted 2007-08-20 (Estimated); Results first posted 2012-03-13 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-02

CONDITIONS: Vascular Disease, Peripheral
Keywords: Restenosis; Superficial Femoral Artery; Prevention of restenosis; Revascularization of the superficial Femoral Artery
MeSH Terms: conditions — Peripheral Vascular Diseases | interventions — Taxes; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- No Drug Treatment Control (No Intervention): Following revascularization, participants did not receive any study drug treatment.
- Proximal to Lesion + IV (Experimental): Participants received an initial intraarterial infusion (proximal to the lesion) of 45 mg/m^2 nanoparticle paclitaxel immediately following revascularization, and a follow-up intravenous injection of 45 mg/m^2 at 7 days.
  Interventions: Drug: Nanoparticle Paclitaxel
- During Flow Arrest (Experimental): Participants received an initial intraarterial infusion (during flow arrest) of 45 mg/m^2 nanoparticle paclitaxel immediately following revascularization.
  Interventions: Drug: Nanoparticle Paclitaxel
- During Flow Arrest + IV (Experimental): Participants received an initial intraarterial infusion (during flow arrest) of 45mg/m^2 nanoparticle paclitaxel immediately following revascularization and a follow-up intravenous injection of 45 mg/m^2 at 7 days.
  Interventions: Drug: Nanoparticle Paclitaxel

INTERVENTIONS:
Drug: Nanoparticle Paclitaxel — Nanoparticle albumin-bound paclitaxel, 45 mg/m^2.
  Other Names: ABI-007; Abraxane®; Coroxane™
  Arms: During Flow Arrest; During Flow Arrest + IV; Proximal to Lesion + IV

SUMMARY:
The purpose of this study is to investigate the prevention of Restenosis following Revascularization of the superficial Femoral Artery (SFA)

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant and non-lactating female and greater than or equal to 18 years of age. All females if child bearing potential must have a negative serum pregnancy test
* Patient is determined to have peripheral artery disease (PAD) classified as Rutherford category 1-4 (grade I/II) - mild, moderate, or severe claudication or ischemic rest pain
* Patient has de novo lesion causing occlusion or an angiographic stenosis of at least 50% in the superficial femoral artery
* Patient has a single or multiple lesions located in the superficial femoral artery with a total length 5-15 cm.
* Normal vessel diameter of the SFA is 4-6 mm
* Patient must have a visibly patent (by angiography) popliteal artery below the target lesion
* No residual flow limiting dissection or residual stenosis greater 30% (visual estimate) after percutaneous balloon angioplasty (PTA) or provisional stenting. Treatment with provisional stenting will be allowed only for flow-limiting dissection, grade C/D or greater than 30 % residual stenosis angiographically after angioplasty alone.
* No target vessel thrombosis confirmed angiography post-PTA procedure
* No distal embolization within target limb
* Patient or his/her legally authorized representative or guardian has been informed about the nature of the study, and has agreed to participate in the study, and signed the Informed Consent Form prior to any premedication, prior to performance of revascularization procedures, and prior to participation in any study-related activities

Exclusion Criteria:

* Women of child bearing potential who do not use adequate contraception
* Patients who have experienced acute onset of claudication
* History of bleeding diathesis, coagulopathy, platelet disorder, or thrombocytopenia
* Patients with lesions requiring treatment with atherectomy or primary stenting
* Target lesion in which PTA failure would require treatment by provisional stenting with more than 2 stents
* Patient has a life expectancy of less than 36 months or there are factors making clinical follow up difficult (no fixed address, etc)
* Additional planned vascular procedure in treated extremity (note that concurrent endovascular treatment of iliac disease is allowable)
* Patient is immunosuppressed or is HIV positive
* Any individual who may refuse a blood transfusion
* Documented major gastrointestinal bleeding within 3 months
* The following lab values at baseline are exclusionary:
* Serum creatinine greater or equal to 2.5 mg/dl
* Platelet count less than 100,000 cells/mm^3
* Uncorrectable coagulopathy with international normalized ratio (INR) greater than 2.0
* Absolute Neutrophil Count (ANC) less than 2000 cells mm^3
* Hemoglobin (Hgb) less than 9 g/dl
* Total Bilirubin greater than 1.5 mg/dl
* Alanine transaminase (SGPT) greater than 2.5 x upper limit normal range (ULN)
* Aspartate transaminase (SGOT) greater than 2.5 x ULN
* Alkaline phosphatase greater than 2.5 x ULN
* Total cholesterol greater than 350 mg/dl or Low Density Lipoprotein greater than 200 mg/dl
* Known allergies/hypersensitivity/contraindication to the study drug, to taxanes, to any required study treatment:aspirin, heparin, clopidogrel bisulfate, stent materials, or to ticlopidine, or dipyridamole
* Patient treated with bivalirudin (Angiomax)
* Pre-existing sensory neuropathy of National Cancer Institute (NCI) Toxicity Grade >1
* Previous participation in another study with any investigational drug or device within the past 30 days or current enrollment in any other clinical protocol or investigational trial
* Renal failure requiring hemodialysis
* Lower extremity or pedal pulse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-01; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: José Iglesias, MD, Study Director — Celgene Corporation
Locations (7):
- United States (7):
  - UC Davis Medical Center, Ellison Ambulatory Care Center Cardiology Suite 3400, Sacramento, California
  - Vascular & Interventional Physicians, Gainsville, Florida
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - Michigan Vascular Research Center, Flint, Michigan
  - Holy Name Hospital, Teaneck, New Jersey
  - Lindner Clinical Trials Center, Cincinnati, Ohio
  - Rhode Island Hospital, Providence, Rhode Island

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Following revascularization, participants did not receive any study drug treatment.
Period: Overall Study
Arm/Group | Control | Proximal to Lesion + IV | During Flow Arrest | During Flow Arrest + IV
Started | 0 | 3 | 1 | 2
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 3 | 1 | 2
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Study Termination | 0 | 2 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Proximal to Lesion + IV | During Flow Arrest | During Flow Arrest + IV | Total
Number analyzed (Participants) | 0 | 3 | 1 | 2 | 6
Age Continuous [Mean (Standard Deviation); unit: years] |  | 69.7 (10.50) | 84.0 (NA) — Standard deviation could not be calculated as only one patient was randomized to this treatment group. | 69.0 (12.73) | 71.8 (10.59)
Gender [Number; unit: participants]
  Female |  | 0 | 0 | 1 | 1
  Male |  | 3 | 1 | 1 | 5
Race/Ethnicity, Customized [Number; unit: participants]
  Asian |  | 0 | 0 | 1 | 1
  White, Non-Hispanic and Non-Latino |  | 3 | 1 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Target Vessel Revascularization at 9 Months
Description: Target vessel revascularization (TVR) was defined as percutaneous revascularization or bypass of the target lesion or any segment of the artery containing the target lesion. The percentage of participants requiring revascularization of the target vessel was determined by stenosis of > 50% confirmed by angiography.
Time Frame: 9 months
Population: Because the study was cancelled after only 6 patients were enrolled, this analysis was not performed.
Measure: Number; unit: percentage of participants
Arm/Group | Control | Proximal to Lesion + IV | During Flow Arrest | During Flow Arrest + IV
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Systolic Velocity Ratio (SVR) > 2.0
Description: The percentage of participants with a systolic velocity ratio > 2.0 assessed using lower extremity arterial duplex ultrasound.
Time Frame: 9 months
Population: Because the study was cancelled after only 6 patients were enrolled, this analysis was not performed.
Measure: Number; unit: percentage of participants
Arm/Group | Control | Proximal to Lesion + IV | During Flow Arrest | During Flow Arrest + IV
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Change From Baseline in Walking Impairment Questionnaire (WIQ) Score
Description: The Walking Impairment Questionnaire (WIQ) is utilized to characterize a patient's walking ability. Scores range from 0 (no difficulty) to 100 (much difficulty).
Time Frame: Baseline and Month 9
Population: Because the study was cancelled after only 6 patients were enrolled, this analysis was not performed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Control | Proximal to Lesion + IV | During Flow Arrest | During Flow Arrest + IV
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Decrease in Ankle Brachial Index (ABI) > 0.15
Description: The percentage of participants with a decrease in the Ankle Brachial Index (ABI) > 0.15.
  Ankle Brachial Index = Systolic Ankle Pressure / Systolic Brachial Pressure.
Time Frame: Baseline and Month 9
Population: Because the study was cancelled after only 6 patients were enrolled, this analysis was not performed.
Measure: Number; unit: percentage of participants
Arm/Group | Control | Proximal to Lesion + IV | During Flow Arrest | During Flow Arrest + IV
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Target Lesion Revascularization (TLR) at 9 Months
Description: Target lesion revascularization (TLR) was defined as repeat percutaneous intervention or bypass surgery of the previously treated target lesion (or blockage). The percentage of participants requiring revascularization of the target lesion was determined by stenosis of > 50% confirmed by angiography.
Time Frame: 9 months
Population: Because the study was cancelled after only 6 patients were enrolled, this analysis was not performed.
Measure: Number; unit: percentage of participants
Arm/Group | Control | Proximal to Lesion + IV | During Flow Arrest | During Flow Arrest + IV
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Deaths
Description: Number of patients who died due to any cause.
Time Frame: Up to 11 months
Population: Treated population.
Measure: Number; unit: participants
Arm/Group | Control | Proximal to Lesion + IV | During Flow Arrest | During Flow Arrest + IV
Number analyzed (Participants) | 0 | 3 | 1 | 2
participants |  | 1 | 0 | 0

7. Secondary Outcome: Number of Participants With Myocardial Infarction (MI)
Description: The number of patients experiencing Myocardial Infarction (MI) during the study. Myocardial Infarction was defined as new pathologic Q waves of at least 0.04 seconds, or an increase in serum creatine kinase to more than twice the normal code together with a pathologic increase in myocardial isoenzymes.
Time Frame: Up to 11 months
Population: Treated population.
Measure: Number; unit: participants
Arm/Group | Control | Proximal to Lesion + IV | During Flow Arrest | During Flow Arrest + IV
Number analyzed (Participants) | 0 | 3 | 1 | 2
participants |  | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With a Stroke
Description: The number of patients experiencing a stroke during the study. Stroke was defined as any sudden development of neurological deficits lasting more than 24 hours, and if a brain imaging study is performed it shows an infarction or hemorrhage. A transient ischemic attack is a neurological deficit lasting less than 24 hours and, if an imaging study is performed, shows no evidence of infarction or hemorrhage.
Time Frame: Up to 11 months
Population: Treated population.
Measure: Number; unit: participants
Arm/Group | Control | Proximal to Lesion + IV | During Flow Arrest | During Flow Arrest + IV
Number analyzed (Participants) | 0 | 3 | 1 | 2
participants |  | 0 | 0 | 0

9. Secondary Outcome: Minimum Lumen Diameter
Description: Minimum lumen diameter (MLD) is defined as the smallest diameter in millimeters (mm) in the arterial segment of interest measured angiographically.
Time Frame: 9 months
Population: Because the study was cancelled after only 6 patients were enrolled, this analysis was not performed.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Control | Proximal to Lesion + IV | During Flow Arrest | During Flow Arrest + IV
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: Late Loss
Description: Late loss is defined as minimum lumen diameter (MLD) immediately post-procedure minus MLD at the time of follow-up, in mm.
Time Frame: Day 1 (following revascularization) and 9 months
Population: Because the study was cancelled after only 6 patients were enrolled, this analysis was not performed.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Control | Proximal to Lesion + IV | During Flow Arrest | During Flow Arrest + IV
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Percentage of Participants With Binary Restenosis
Description: Binary restenosis was defined by a >50% diameter stenosis at follow-up study, assessed by angiography.
Time Frame: 9 months
Population: Because the study was cancelled after only 6 patients were enrolled, this analysis was not performed.
Measure: Number; unit: percentage of participants
Arm/Group | Control | Proximal to Lesion + IV | During Flow Arrest | During Flow Arrest + IV
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Secondary Outcome: Diameter Stenosis
Description: Diameter stenosis is calculated as [1 - (minimum lumen diameter (MLD) / reference vessel diameter)] * 100, where the reference vessel diameter is the vessel diameter measured in a healthy segment of the target vessel proximal as close as possible to the lesion.
Time Frame: 9 months
Population: Because the study was cancelled after only 6 patients were enrolled, this analysis was not performed.
Measure: Mean (Standard Deviation); unit: percent diameter stenosis
Arm/Group | Control | Proximal to Lesion + IV | During Flow Arrest | During Flow Arrest + IV
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 11 months
Arm/Group | Control | Proximal to Lesion + IV | During Flow Arrest | During Flow Arrest + IV
Serious Adverse Events (participants affected / at risk) | 0/0 | 1/3 | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/0 | 1/3 | 0/1 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=0) | Proximal to Lesion + IV (N=3) | During Flow Arrest (N=1) | During Flow Arrest + IV (N=2)
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=0) | Proximal to Lesion + IV (N=3) | During Flow Arrest (N=1) | During Flow Arrest + IV (N=2)
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pain in extremity (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
* Study data will not be published in part before complete multicenter data have been reported in full, unless more than 18 months have elapsed since completion of the Study.
* Investigator/institution must supply copy of presentation or publication to Celgene 30 days of prior to submission for publication. Celgene may request in writing within that 30 days that Celgene Confidential Information be deleted or be granted a 60 day delay prior to publication for intellectual property filings.